CLINICAL TRIAL: NCT00345579
Title: A Single-blind, Randomized, Controlled, Multinational Study for the Evaluation of Safety of GlaxoSmithKline (GSK) Biologicals' Investigational Vaccination Regimen Compared to Monovalent Haemophilus Influenzae Type b (Hib) Control Vaccine in Healthy Infants at 2, 4, 6, and 12 to 15 Months of Age.
Brief Title: Safety of Hib-MenCY-TT Vaccine Versus Licensed Hib Conjugate Vaccine, Given at 2, 4, 6 and 12 to 15 Months of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 105987
Record Dates: First submitted 2006-06-26; First posted 2006-06-28 (Estimated); Results first posted 2012-07-20 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-11

CONDITIONS: Haemophilus Influenzae Type b; Neisseria Meningitidis
Keywords: Prophylaxis; Neisseria meningitidis Vaccines, conjugate; Infants; Meningococcal vaccines; H. influenzae type B vaccine; Humans; Safety
MeSH Terms: conditions — Haemophilus Infections | interventions — Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate; PEDIARIX

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Menhibrix Group (Experimental): Subjects received 3 doses of Menhibrix vaccine (at 2, 4 and 6 months of age, study Months 0, 2 and 4), co-administered with Pediarix/Infanrix penta as a primary vaccination course and a fourth dose of Menhibrix vaccine at 12-15 months of age in the study NCT00345683. Menhibrix was administered intramuscularly in the upper right thigh and co-administered Pediarix/Infanrix penta vaccine was injected intramuscularly in the upper left thigh.
  Interventions: Biological: GSK Biologicals' Haemophilus influenzae type b and Neisseria meningitidis serogroups C and Y-tetanus toxoid conjugate vaccine combined 792014; Biological: Pediarix/Infanrix Penta
- ActHIB Group (Active Comparator): Subjects received 3 doses of ActHIB vaccine (at 2, 4 and 6 months of age, study Months 0, 2 and 4), co-administered with Pediarix/Infanrix penta as a primary vaccination course and 1 dose of PedvaxHib vaccine as a booster at 12-15 months of age in the study NCT00345683. ActHIB and PedvaxHib vaccines were administered intramuscularly in the upper right thigh and co-administered Pediarix/Infanrix penta vaccine was injected intramuscularly in the upper left thigh.
  Interventions: Biological: ActHIB; Biological: Pediarix/Infanrix Penta

INTERVENTIONS:
Biological: GSK Biologicals' Haemophilus influenzae type b and Neisseria meningitidis serogroups C and Y-tetanus toxoid conjugate vaccine combined 792014 — 3-dose intramuscular injection
  Arms: Menhibrix Group
Biological: ActHIB — 3-dose intramuscular injection
  Arms: ActHIB Group
Biological: Pediarix/Infanrix Penta — 3-dose intramuscular injection

SUMMARY:
The primary phase of this study is evaluating the safety of Hib-MenCY-TT vaccine compared to a control group receiving licensed Hib conjugate vaccine, when each are co-administered with Pediarix® to healthy infants at 2, 4, and 6 months of age.

This protocol posting deals with objectives & outcome measures of the primary phase of the study. The objectives & outcome measures of the Booster phase are presented in a separate protocol posting (NCT number = 00345683).

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007

DETAILED DESCRIPTION:
Pediarix/Infanrix Penta and Prevnar should be co-administered to all subjects in all study groups according to a 2, 4, and 6 month schedule concomitantly with study vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Subjects for whom the investigator believes that parents/guardians can and will comply with the requirements of the protocol.
* A male or female between, and including, 6 and 12 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born after 36 weeks gestation.
* Infants who have not received a previous dose of hepatitis B vaccine or those who have received only 1 dose of hepatitis B vaccine administered at least 30 days prior to enrolment.
* Infants may have received a birth dose of Bacillus Calmette-Guérin (BCG) vaccine.

Exclusion criteria:

Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.

* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of study vaccine(s).
* Previous vaccination against Neisseria meningitidis, Haemophilus influenzae type b, diphtheria, tetanus, pertussis, and/or poliovirus; more than one previous dose of hepatitis B vaccine.
* In country(ies) where Prevnar will be provided by GSK Biologicals, previous vaccination with Prevnar.
* History of Neisseria meningitidis, Haemophilus influenzae type b, diphtheria, tetanus, pertussis, hepatitis B, and/or poliovirus disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, including dry natural latex rubber.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at time of enrollment.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Concurrent participation in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4432 (Actual)
Dates: Start 2006-09; Primary Completion 2007-10 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (55):
- United States (54):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Benton, Arkansas
  - GSK Investigational Site, Fayetteville, Arkansas
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Madera, California
  - GSK Investigational Site, Slinas, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, Boulder, Colorado
  - GSK Investigational Site, Longmont, Colorado
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Oak Lawn, Illinois
  - GSK Investigational Site, Waukee, Iowa
  - GSK Investigational Site, West Desmoines, Iowa
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Bossier City, Louisiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Jamaica Plain, Massachusetts
  - GSK Investigational Site, Nies, Michigan
  - GSK Investigational Site, Portage, Michigan
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, New Hartford, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Clyde, North Carolina
  - GSK Investigational Site, Deerfield, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Sylva, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, North Canton, Ohio
  - GSK Investigational Site, South Euclid, Ohio
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Wexford, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Katy, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, Orem, Utah
  - GSK Investigational Site, Pleasant Gorve, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Marshfield, Wisconsin
- GSK Investigational Site, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bryant KA, Marshall GS. Haemophilus influenzae type b-Neisseria meningitidis serogroups C and Y tetanus toxoid conjugate vaccine for infants and toddlers. Expert Rev Vaccines. 2011 Jul;10(7):941-50. doi: 10.1586/erv.11.90. PMID 21806393
- [Background] Rinderknecht S, Bryant K, Nolan T, Pavia-Ruz N, Doniz CA, Weber MA, Cohen C, Aris E, Mesaros N, Miller JM. The safety profile of Haemophilus influenzae type b-Neisseria meningitidis serogroups C and Y tetanus toxoid conjugate vaccine (HibMenCY). Hum Vaccin Immunother. 2012 Mar;8(3):304-11. doi: 10.4161/hv.18752. Epub 2012 Feb 13. PMID 22327493
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 105987 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 105987 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 105987 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 105987 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 105987 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 105987 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This summary presents results for the primary vaccination phase up to the end of the extended safety follow-up (until, but excluding, the booster dose at 12-15 months of age). For results about the booster/fourth dose phase, see study NCT00345683.
Pre-assignment Details: Of the 4432 subjects enrolled, 4391 were vaccinated and 4162 completed the primary vaccination phase of the study (3114 in the MenHibrix Group and 1048 in the ActHIB Group).
Period: Overall Study
Arm/Group | MenHibrix Group | ActHIB Group
Started | 3278 | 1113
Completed | 3114 | 1048
Not Completed | 164 | 65
Not completed — Adverse Event | 9 | 6
Not completed — Protocol Violation | 14 | 5
Not completed — Withdrawal by Subject | 50 | 17
Not completed — Lost to Follow-up | 82 | 36
Not completed — Other | 9 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MenHibrix Group | ActHIB Group | Total
Number analyzed (Participants) | 3278 | 1113 | 4391
Age, Continuous [Mean (Standard Deviation); unit: Days] | 58.6 (10.45) | 59.0 (10.39) | 58.8 (10.42)
Gender [Count of Participants; unit: Participants]
  Female | 1576 | 557 | 2133
  Male | 1702 | 556 | 2258

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Time Frame: From Dose 1 up to Day 30 after Dose 3 (from study Month 0 up to study Month 5)
Population: The Primary Total Vaccinated cohort included all subjects with at least one primary vaccine dose of study vaccine administered.
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 3278 | 1113
Subjects | 109 | 33

2. Primary Outcome: Number of Subjects Reporting New Onset of Chronic Illnesses (NOCIs)
Description: NOCIs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: From Dose 1 up to Day 30 after Dose 3 (from study Month 0 up to study Month 5)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 3278 | 1113
Subjects | 50 | 18

3. Primary Outcome: Number of Subjects Reporting Rash
Description: Rash assessed was hives, idiopathic thrombocytopenic purpura, petechiae.
Time Frame: From Dose 1 up to Day 30 after Dose 3 (from study Month 0 up to study Month 5)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 3278 | 1113
Subjects | 243 | 81

4. Primary Outcome: Number of Subjects Reporting Adverse Events Resulting in Emergency Room (ER)
Time Frame: From Dose 1 up to Day 30 after Dose 3 (from study Month 0 up to study Month 5)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 3278 | 1113
Subjects | 114 | 44

5. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 1
Time Frame: From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 3278 | 1113
Subjects | 157 | 48

6. Primary Outcome: Number of Subjects With New Onset of Chronic Illnesses (NOCIs)
Description: NOCIs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 3278 | 1113
Subjects | 66 | 25

7. Primary Outcome: Number of Subjects With Rash
Description: Rash assessed was hives, idiopathic thrombocytopenic purpura, petechiae
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 3278 | 1113
Subjects | 386 | 134

8. Primary Outcome: Number of Subjects With Adverse Events Resulting in Emergency Room (ER)
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Number; unit: Subjects
Groups:
- MenHibrix Group: Subjects received 3 doses of MenHibrix vaccine (at 2, 4 and 6 months of age, study Months 0, 2 and 4), co-administered with Pediarix/Infanrix penta as a primary vaccination course and a fourth dose of MenHibrix vaccine at 12-15 months of age in the study NCT00345683. MenHhibrix was administered intramuscularly in the upper right thigh and co-administered Pediarix/Infanrix penta vaccine was injected intramuscularly in the upper left thigh.
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 3278 | 1113
Subjects | 198 | 69

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Description: Solicited symptoms and unsolicited AEs were not collected during the study. Only information about specific categories of AEs (SAEs, NOCIs, rash and AEs resulting in ER visits) were collected in this study.
Arm/Group | MenHibrix Group | ActHIB Group
Serious Adverse Events (participants affected / at risk) | 157/3278 | 48/1113
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MenHibrix Group (N=3278) | ActHIB Group (N=1113)
Febrile convulsion (Nervous system disorders) | 5 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Fractured skull depressed (Injury, poisoning and procedural complications) | 0 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Haematoma (Vascular disorders) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Haematuria (Renal and urinary disorders) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Haemorrhagic infarction (Vascular disorders) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Ileus (Gastrointestinal disorders) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Oedema peripheral (General disorders) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Perirectal abscess (Infections and infestations) | 0 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Septic shock (Infections and infestations) | 0 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Varicella (Infections and infestations) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Gastroenteritis (Infections and infestations) | 32 | 11 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Bronchiolitis (Infections and infestations) | 39 | 6 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Bronchopneumonia (Infections and infestations) | 17 | 9 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Dehydration (Metabolism and nutrition disorders) | 5 | 5 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Pneumonia (Infections and infestations) | 9 | 2 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 10 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Viral infection (Infections and infestations) | 0 | 2 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Gastroenteritis rotavirus (Infections and infestations) | 2 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Otitis media (Infections and infestations) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Urinary tract infection (Infections and infestations) | 4 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Head injury (Injury, poisoning and procedural complications) | 9 | 2 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Pyrexia (General disorders) | 1 | 2 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 3 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Croup infectious (Infections and infestations) | 2 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Intussusception (Gastrointestinal disorders) | 0 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Sudden infant death syndrome (General disorders) | 3 | 2 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Upper respiratory tract infection (Infections and infestations) | 1 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Pyelonephritis (Infections and infestations) | 3 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Vomiting (Gastrointestinal disorders) | 0 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Cellulitis (Infections and infestations) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Convulsion (Nervous system disorders) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Pharyngitis (Infections and infestations) | 2 | 2 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Gastroenteritis viral (Infections and infestations) | 1 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Skull fracture (Injury, poisoning and procedural complications) | 3 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Tracheitis (Infections and infestations) | 1 | 2 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Hypovolaemic shock (Vascular disorders) | 2 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Influenza (Infections and infestations) | 0 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Lobar pneumonia (Infections and infestations) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Nasopharyngitis (Infections and infestations) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Nystagmus (Nervous system disorders) | 1 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Subcutaneous abscess (Infections and infestations) | 2 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Abdominal distension (Gastrointestinal disorders) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Anaphylactic reaction (Immune system disorders) | 0 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Breath holding (Psychiatric disorders) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Bronchitis (Infections and infestations) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Cardiac failure congestive (Cardiac disorders) | 0 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Child abuse (Social circumstances) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Constipation (Gastrointestinal disorders) | 0 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Depressed level of consciousness (Nervous system disorders) | 0 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Epilepsy (Nervous system disorders) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Eye injury (Injury, poisoning and procedural complications) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Skin injury (Injury, poisoning and procedural complications) | 1 | 0 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)
Tonsillitis (Infections and infestations) | 0 | 1 — From Dose 1 through but excluding the fourth dose (from study Month 0 up to the booster vaccination at 12-15 months of age)

LIMITATIONS AND CAVEATS:
Solicited symptoms and unslocited AEs were not collected during this study. Only information about specific categories of AEs (SAEs, NOCIs, rash and AEs resulting in ER visits) were collected in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.